CLINICAL TRIAL: NCT01919177
Title: Effect of Inorganic Nitrates on Arterial Hemodynamics and Exercise Capacity
Brief Title: Effect of Inorganic Nitrates (Beetroot Juice) on Arterial Hemodynamics and Exercise Capacity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Corporal Michael J. Crescenz VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Julio A.Chirinos, Director of non-invasive imaging & Assistant Professor of Medicine, Corporal Michael J. Crescenz VA Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01415
Record Dates: First submitted 2013-07-22; First posted 2013-08-08 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Heart Failure With Normal Ejection Fraction
Keywords: Heart Failure; Arterial hemodynamics; Exercise capacity; Mitochondrial oxidative capacity
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nitrate rich beetroot juice (Active Comparator): Subjects with heart failure with preserved ejection fraction will receive 140 mL of Nitrate-rich concentrated beetroot juice (containing 12 mmol of NO-3). This will be a cross-over study. Therefore all subjects will receive both interventions, but the order of the interventions will be randomized.
  Interventions: Dietary Supplement: Nitrate rich beetroot juice
- Nitrate depleted beetroot juice (Placebo Comparator): Subjects with heart failure with preserved ejection fraction will receive 140 mL of nitrate-depleted beetroot juice (containing <0.01 mmol of NO-3).This will be a cross-over study. Therefore all subjects will receive both interventions, but the order of the interventions will be randomized.
  Interventions: Dietary Supplement: Nitrate depleted beetroot juice

INTERVENTIONS:
Dietary Supplement: Nitrate rich beetroot juice — Subjects will receive 140 mL of Nitrate-rich concentrated beetroot juice.
  Other Names: Beet It Stamina Sports shots
  Arms: Nitrate rich beetroot juice
Dietary Supplement: Nitrate depleted beetroot juice — Subjects will receive 140 mL of nitrate-depleted beetroot juice.
  Other Names: Beet It nitrate extracted (depleted) placebo shots
  Arms: Nitrate depleted beetroot juice

SUMMARY:
The main objective is to test the hypothesis that inorganic nitrate supplementation will: (1) Improve exercise efficiency and performance; (2) Enhance the systemic vasodilator reserve during exercise and specifically, the vasodilator response in exercising muscle; (3) Reduce arterial wave reflections and arterial load; (4) Improve skeletal muscle mitochondrial function in subjects with heart failure with preserved ejection fraction.

DETAILED DESCRIPTION:
This represents a series of double-blind, controlled pilot randomized studies in which the effects of nitrate-rich beetroot juice and nitrate-depleted beetroot juice will be assessed in patients with heart failure and preserved ejection fraction (n=20). A total of 20 subjects will be enrolled over a 1.5 year period and randomized in a cross-over design to a single dose of nitrate-rich beetroot juice and nitrate-depleted beetroot juice. The order of the interventions will be randomized; thus, all subjects will receive the nitrate-rich and nitrate-depleted juice, with a 4-7 day washout period in-between studies.

ELIGIBILITY:
Inclusion Criteria:

The investigators will enroll 20 subjects >18 years of age who have a diagnosis of heart failure with preserved ejection fraction (>50%) by 2d echocardiography, with current New York Heart Association Class II-IV symptoms.

In addition, subjects with heart failure must meet the following inclusion criteria:

1. Chronic treatment with a loop diuretic for control of HF symptoms.
2. If EF is normal, subjects must demonstrate elevated filling pressures as evidenced by at least one of the following: a) left atrial enlargement (LAVI > 32 mL/m2); b) at least stage II diastolic dysfunction; c) Documentation of elevated NT-pro BNP levels or other natriuretic peptide marker (BNP, ANP) according to the laboratory and assay upper limit of normal in the previous year.
3. Stable medical therapy as defined by: (I) No addition or removal of ACE, ARB, beta-blockers, or calcium channel blockers (CCBs) for 30 days. (II) No change in dosage of ACE, ARBs, beta-blockers or CCBs of more than 100% for 30 days. (III) No change in diuretic dose for 10 days.

Exclusion Criteria:

1. Rhythm other than sinus rhythm (i.e., atrial fibrillation).
2. Neuromuscular, orthopedic or other non-cardiac condition that prevents patient from exercising.
3. Valve disease (> mild aortic or mitral stenosis; > moderate aortic or mitral regurgitation).
4. Hypertrophic cardiomyopathy.
5. Known infiltrative or inflammatory myocardial disease (amyloid, sarcoid).
6. Pericardial disease.
7. Primary pulmonary arteriopathy.
8. Have experienced a myocardial infarction or unstable angina, or have undergone percutaneous transluminal coronary angiography (PTCA) or coronary artery bypass grafting (CABG) within 60 days prior to consent, or requires either PTCA or CABG at the time of consent.
9. Other clinically important causes of dyspnea such as morbid obesity or significant lung disease defined by clinical judgment or use of steroids or oxygen for lung disease within the past 6 months.
10. Systolic blood pressure < 110 mmHg or > 180 mm Hg.
11. Diastolic blood pressure < 40 mmHg or > 100 mmHg.
12. Resting heart rate (HR) > 100 bpm.
13. Hemoglobin <10 g/dL.
14. Patients with known severe liver disease (AST > 3x normal, alkaline phosphatase or bilirubin > 2x normal).
15. Patients with a clinically indicated stress test demonstrating significant ischemia within a year of enrollment which was not followed by percutaneous or surgical revascularization.
16. Current therapy with phosphodiesterase inhibitors, such as sildenafil, vardanafil or tadalafil.
17. Known allergies to beetroot or lemon juice.
18. Current use of organic nitrates or phosphodiesterase inhibitors.
19. Pregnancy. Although beetroot juice has not knows teratogenic effects, we feel that not enough data exist in this regard. Therefore, all females patients of reproductive age will be required to undergo a pregnancy test prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-01; Primary Completion 2014-09 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in Peak exercise efficiency during maximal effort supine-bicycle exercise and peak oxygen consumption (VO2) during a maximal effort supine-bicycle exercise test | Baseline study, repeat study 4-7 days later
  We will assess the relationship between total power output and total O2 consumption (VO2, assessed via expired gas analysis) during a maximal-effort supine bicycle exercise test.

SECONDARY OUTCOMES:
Change in Arterial wave reflection magnitude | Baseline study, repeat study 4-7 days later
  Reflection wave magnitude will be assessed using arterial tonometry to arrive at the augmentation index. The data will also be processed using custom designed software for wave separation analysis to quantify the magnitude and timing of the reflected waves.
Change in Peripheral vascular resistance, total arterial compliance and reflection magnitude during supine bicycle peak exercise | Baseline study, repeat study 4-7 days later
Change in lower extremity exercise vasodilator reserve (change in femoral vascular resistance between rest and maximal effort supine-bicycle exercise) | Baseline study, repeat study 4-7 days later
Change in lower extremity blood flow reserve (change in femoral artery blood flow between rest and maximal effort supine-bicycle exercise) | Baseline study, repeat study 4-7 days later
Change in submaximal exercise efficiency (O2 consumption per power output during submaximal exercise and standardized handgrip exercise) | Baseline study, repeat study 4-7 days later
Change in Skeletal Muscle Mitochondrial Oxidative Capacity | Baseline study, repeat study 4-7 days later
  The investigators will assess the oxygen consumption recovery kinetics after moderate forearm exercise, using repeated cuff brachial artery occlusions and near-infrared spectroscopy.
Change in post-ischemic vasodilatory response | Baseline study, repeat study 4-7 days later
  The investigators will assess the post-ischemic vasodilatory response in the forearm using brachial artery pulsed wave Doppler interrogations before and after inflation of a brachial cuff at 200 mmHg for 5 minutes. The investigators will also assess forearm microvascular skeletal muscle flow with near-infrared spectroscopy and forearm skin microvascular flow using laser Doppler.

CONTACTS AND LOCATIONS:
Overall Officials: Julio A Chirinos, MD, PhD, Principal Investigator — Philadelphia VA Medical Center & University of Pennsylvania
Locations (1):
- Philadelphia Veterans Affairs Medical Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] American Thoracic Society; American College of Chest Physicians. ATS/ACCP Statement on cardiopulmonary exercise testing. Am J Respir Crit Care Med. 2003 Jan 15;167(2):211-77. doi: 10.1164/rccm.167.2.211. No abstract available. PMID 12524257
- [Background] Manetos C, Dimopoulos S, Tzanis G, Vakrou S, Tasoulis A, Kapelios C, Agapitou V, Ntalianis A, Terrovitis J, Nanas S. Skeletal muscle microcirculatory abnormalities are associated with exercise intolerance, ventilatory inefficiency, and impaired autonomic control in heart failure. J Heart Lung Transplant. 2011 Dec;30(12):1403-8. doi: 10.1016/j.healun.2011.08.020. Epub 2011 Oct 7. PMID 21982360
- [Result] Zamani P, Rawat D, Shiva-Kumar P, Geraci S, Bhuva R, Konda P, Doulias PT, Ischiropoulos H, Townsend RR, Margulies KB, Cappola TP, Poole DC, Chirinos JA. Effect of inorganic nitrate on exercise capacity in heart failure with preserved ejection fraction. Circulation. 2015 Jan 27;131(4):371-80; discussion 380. doi: 10.1161/CIRCULATIONAHA.114.012957. Epub 2014 Dec 22. PMID 25533966